CLINICAL TRIAL: NCT05862376
Title: Nutritional Status and Iodized Salt Use Among School-aged Children Living in Phu Kut City, Xieng Khouang Province, Lao PDR
Brief Title: Nutritional Status and Iodized Salt Use Among School-aged Children
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 067/NECHR
Record Dates: First submitted 2023-04-27; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Iodine Deficiency
Keywords: Nutritional status; Iodized salt; School-aged children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine and explore the iodized salt concentration provided in the local community, especially in the Phu Kut district whether it meets the standard or not. This district is located in a mountainous area which means that the local community confronts with geographical access due to the limited transportation and road condition, in addition, it is quite far from downtown approximately 26 kilometers and it is difficult to access the iodized salt consumption.

On the other hand, since 2013, the Lao People's Democratic Republic has implemented the iodized survey of urine among the primary students, this time could be the chance to compare based on the previous data, which will be an important source of the data for certifying the quality of iodized salt available in the local community that could be one cause of lacking iodized salt intake. Furthermore, the investigators could conduct the survey and monitor the current action plan related to iodized consumption in Laos as well, in order to eradicate diseases concerning with lacking iodized salt intake.

Objectives

1. To investigate the nutritional status of school-aged children (SAC) living in Phu Kut City, Xieng Khouang province.
2. To investigate the iodine status and iodized salt use of school-aged children (SAC) living in Phu Kut City, Xieng Khouang province.

DETAILED DESCRIPTION:
Malnutrition Situation in Lao PDR. The Lao PDR has witnessed significant improvements in its Gross Domestic Product (GDP) for the past 2 decades. However, this does not commensurate with reductions in food insecurity and malnutrition (NNS, 2016). There exist significant disparities in income and living conditions between the rich and the poor; rural and urban dwellers; literates and illiterates (MOH-Lao PDR, 2014).

Lao PDR has the highest prevalence of stunting in the ASEAN region with an estimated 33% of children under 5 years being too short for their age (stunted) and 9.6% acutely malnourished (LSIS, 2017). Whilst recognizing the marginal reductions in the prevalence of malnutrition, the rates are relatively higher than recommended thresholds and of public health significance.

Micronutrient deficiency among the population is at an alarming level and calls for urgent action. 2 out of 5 children under 5 years are anemic and another 30% of preschool children are suffering from Vitamin A Deficiency (VAD). 36.2% of women in reproductive age are anemic with less than 20% of the general population consuming adequately iodized salt (LSIS, 2011-2012). In 2017, it can be seen that in the whole country, there are households that consume iodized salt increased to 89.2%, specifically in Xieng Khouang province it is 87.6% (LSIS, 2017).

Most recently in 2018, according to the monitoring report on the quality of iodized salt of the Department of Food and Drug, the Ministry of Health conducted a survey to check the quality of iodized salt in 8 provinces: Vientian capital (Vernkham salt factory), Vientiane province (Ban Bor salt factory), Lung Namtha province (Boten salt factory), Oudomxay province (Elephant brand salt factory), Borikhamxay (Song Kone Salt factory), Savannakhet (Natei Salt factory, Kasay Salt factory and Kasay Thip salt factory), Xieng Khouang province and Huaphan province (imported salt, market salt and household salt). This report found that only 2 out of 9 salt factories produced iodized salt according to the standard (40 ppm -60 ppm) namely Vern Kham Salt Factory and Salt Factory, almost 80% of factory machinery is dilapidated, lack of improvement, looking for spare parts for injectors, there is no place to sell them, lack of mixing techniques and iodine is expensive.

In the Xieng Khouang province, there is no any iodized salt factory, the local people just consumed the imported products. but they could detect the iodized salt concentration selling in the market and in the household. The results from iodized salt testing from 5 target districts have been done from the sampling in the district for a total of 125 samples from 10 trade names of the iodized salt. Unfortunately, there is no iodized salt trade name that meets the standard. Referring to the detail of the trade name and results of iodized salt testing below from five target districts:

No Iodized salt brand name Factory Iodine content (ppm)

1. Iodize salt (spoon tradename) Koksaath 34.8
2. Iodize salt (spoon tradename) Koksaath 23.8
3. Iodize salt (spoon tradename) Koksaath 26.7
4. Iodize salt (spoon tradename) Koksaath 1
5. Iodize salt (carriage tradename) Vernkham 19.4
6. Iodize salt (carriage tradename) Vernkham 22.5
7. Iodize salt (carriage tradename) Vernkham 24.1
8. Muối i ốt (Female tradename) Vietnam iodize salt 1
9. Muối i ốt (Female tradename) Vietnam iodize salt 3.4
10. Muối i ốt (Female tradename) Vietnam iodize salt 2.3

To determine and explore the iodized salt concentration provided in the local community, especially in the Phu Kut district whether it meets the standard or not. This district is located in a mountainous area which means that the local community confronts with geographical access due to the limited transportation and road condition, in addition, it is quite far from downtown approximately 26 kilometers and it is difficult to access the iodized salt consumption.

On the other hand, since 2013, the Lao People's Democratic Republic has implemented the iodized survey of urine among the primary students, this time could be the chance to compare based on the previous data, which will be an important source of the data for certifying the quality of iodized salt available in the local community that could be one cause of lacking iodized salt intake. Furthermore, the investigators could conduct the survey and monitor the current action plan related to iodized consumption in Laos as well, in order to eradicate diseases concerning with lacking of iodized salt intake.

Objectives

1. To investigate the nutritional status of school-aged children (SAC) living in Phu Kut city, Xieng Khouang province.
2. To investigate the iodine status and iodized salt use of school-aged children (SAC) living in Phu Kut city, Xieng Khouang province.

ELIGIBILITY:
Inclusion Criteria:

* School-aged children aged 6-12 year olds and their parents who living in Phu Kut city, Xieng Khouang province.

Exclusion Criteria:

* Inability to understand the information sheet and the informed consent form due to cognitive or language reasons

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School-aged children aged 6-12 year olds and their parents who living in Phu Kut city, Xieng Khouang province.
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Iodine status | 1 year
  Median iodine urinary concentration of school-age children (cut-off values for urinary iodine; deficiency, iodine urinary concentration <100 ug/L, adequate, iodine urinary concentration 100 -199 ug/L, above requirement, iodine urinary concentration 200-299 ug/L, excessive, iodine urinary concentration ≥300).

SECONDARY OUTCOMES:
iodized salt use | 1 year
  Iodine content in salt samples was analyzed by iodometric titration in the analytical room.

CONTACTS AND LOCATIONS:
Overall Officials: Khouanheuane Sengkhamyong, PhD., Principal Investigator — Vientiane, Lao PDR
Locations (2):
- Thailand (2):
  - Institute of Nutrition Mahidol University, Salaya, Changwat Nakhon Pathom
  - Institute of Nutrition, Salaya, Changwat Nakhon Pathom

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] IFPRI. Global Nutrition Report 2016: From Promise to Impact: Ending Malnutrition by 2030. International Food Policy Research Institute, 2016 Washington, DC.
- [Background] McGuire S. International Food Policy Research Institute. 2014. Washington, DC: Global Nutrition Report 2014: actions and accountability to accelerate the world's progress on nutrition. Adv Nutr. 2015 May 15;6(3):278-9. doi: 10.3945/an.115.008599. Print 2015 May. No abstract available. PMID 25979494
- [Background] Hilal E. Nutrition, human rights, and the SDGs-21st Century Global Dynamics. Global-e 2016; Vol 9, Issue 11.
- [Background] UNICEF. State of the world's children: A fair chance for every child, UNICEF, 2016 New York.
- [Background] ASEAN/UNICEF/WHO. Regional Report on Nutrition Security in ASEAN, 2016 Volume 2. Bangkok; UNICEF.
- [Background] Government of Lao PDR. National Nutrition Strategy and Plan of Action 2016-2020 (NNSPA, 2016-2020). 2015.
- [Background] Ministry of Health & Lao Statistical Bureau. Lao Social Indicator Survey (LSIS) 2011 - 12 (Multiple Indicator Cluster Survey / Demographic and Health Survey), December 2012.
- [Background] Ministry of Health & Lao Statistical Bureau. Lao Social Indicator Survey (LSIS) 2017 (Multiple Indicator Cluster Survey / Demographic and Health Survey). 2018.
- [Background] National strategy on Nutrition 2025 and Plan of Action 2016-2020, Lao PDR.
- [Background] WHO Growth reference data for 5-19 years, 2007. Available at: https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators.
- [Background] The International Council for Control of Iodine Deficiency Disorders (ICCIDD), 1995, Monitoring Universal Salt Iodization Programmes, January 1995, pp. 86-101.
- [Background] Pino S, Fang SL, Braverman LE. Ammonium persulfate: a safe alternative oxidizing reagent for measuring urinary iodine. Clin Chem. 1996 Feb;42(2):239-43. PMID 8595717
- [Background] Country Nutrition Profiles: Lao PDR. Global Nutrition Report 2021. Available at: https://globalnutritionreport.org/resources/nutrition-profiles/asia/south-eastern-asia/lao-peoples-democratic-republic/.